CLINICAL TRIAL: NCT02503371
Title: The Effect of In Vitro Fertilization on Coagulation Parameters as Measured by Thromboelastogram
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharonorbach, Dr. Sharon Orbach, Rabin Medical Center
Other Study IDs: 0332-11-RMC
Record Dates: First submitted 2015-07-12; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Fertilization in Vitro and Blood Coagulation Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women under IVF stimulation at the begining and end: Coagulation parameters will be measured for all parturients at the beginning and conclusion of an IVF simulation cycle with the use of thromboelastogram
  Interventions: Other: Blood coagulation anyalsis by Thromboelastogram

INTERVENTIONS:
Other: Blood coagulation anyalsis by Thromboelastogram — Two blood tests will be taken during routine tests from all parturient s undergoing IVF treatment before starting gonadotropins treatment (the first few days of menstruation) and at the height of hormone therapy prior to egg retrieval Coagulation parameters will be measured by the use of Thromboelastogram

SUMMARY:
Since its introduction in 1978, over 3.75 million babies have been born using in vitro fertilization (IVF). Maturing ovarian follicles lead to a large rise in estrogen to supra-physiological levels . This increase in estrogen has been shown to cause a hypercoagulable state, leading at times to arterial and venous thrombosis.(Thromboelastogram (TEG) is a point of care whole blood hemostatsis analyzer mimicking in vivo conditions and measuring visco elastic properties of the clot. The TEG shows effect of most of the components of hemostatsis: coagulation factors, fibrinogen, platelets and fibrinolysis. Components of TEG include R, reflecting coagulation factor cascade, alpha angle and K measurements reflecting fibrin function, MA reflecting mostly thrombocyte function, coagulation index (CI) measuring global hemostatic statis and LY30 measuring fibrinolysis.

In this study the investigators would like to measure serum estrogen levels and (TEG) in parturients at the beginning and conclusion of an IVF simulation cycle and evaluate how it's influnence on coagulation parameters, and wheather or not a large sample size will effect primary outcomes.

Secondarily the investigators would like to see if estrogen levels are predictors of coagulation parameters and see if age influences TEG parameters

ELIGIBILITY:
Inclusion Criteria:

* Parturients above 18 undergoing in-vitro fertilization at rabin medical center, with the ability to comply with the study requriments.

Exclusion Criteria:

Parturients were excluded if they had;

* hypertension,
* diabetes,
* anticoagulation therapy or any platelet disorder,
* or were not able to comply with study requirments.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parturients undergoing in-vitro fertilization treatment
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Measurement of fibrin function in parturients undergoing IVF by Thromboelastogram | one year
Measurement of thrombocyte function in parturients undergoing IVF by Thromboelastogram | one year
Measurement of global hemostatic statis in parturients undergoing IVF by Thromboelastogram | one year
Measurement of fibrinolysisin parturients undergoing IVF by Thromboelastogram | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel